CLINICAL TRIAL: NCT01089413
Title: A Multicenter, Non-interventional, Post-authorization Study to Observe in Daily Clinical Practice the Treatment Duration of Patients Treated With Avastin (Bevacizumab) in 1st Line mCRC in Belgium
Brief Title: Observational Study of Bevacizumab [Avastin] in Patients With Metastatic Colorectal Cancer (AVASTART)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25117
Record Dates: First submitted 2010-03-15; First posted 2010-03-18 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Drug: bevacizumab [Avastin]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — As prescribed by physician

SUMMARY:
This observational study will assess the treatment duration, progression-free survival, reason for stopping treatment and patient and tumor characteristics of bevacizumab [Avastin] treatment in patients with metastatic colorectal cancer. Data will be collected for approximately 34 months. The target sample size is >300 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients =/<18 years of age
* metastatic colorectal cancer
* patients for whom the physician has prescribed bevacizumab [Avastin] for the treatment of 1st line metastatic colorectal cancer
* patients, who have given written informed consent

Exclusion Criteria:

* hypersensitivity to recombinant human or humanised antibodies
* pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 1st line treatment with bevacizumab in Belgium
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Belgium (19):
  - Aalst
  - Antwerp
  - Assebroek
  - Aye
  - Bruges
  - Brussels
  - Charleroi
  - Haine-Saint-Paul
  - Hasselt
  - Ieper
  - Kortrijk
  - Liège
  - Mons
  - Namur
  - Roeselare
  - Sint-Niklaas
  - Tongeren
  - Tournai
  - Vilvoorde

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Overall: All participants with Metastatic Colorectal Cancer (mCRC) for whom the physician decided to prescribe bevacizumab (Avastin) as part of their first line treatment and in line with current Summary of Product Characteristics (SmPC) (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
Period: Overall Study
Arm/Group | Bevacizumab: Overall
Started | 201
Received Bevacizumab in First Line | 199
Completed | 0
Not Completed | 201
Not completed — Lost to Follow-up | 1
Not completed — Progressive Disease | 93
Not completed — Participant Withdrew Consent | 1
Not completed — Unacceptable Toxicity | 12
Not completed — Death | 10
Not completed — Metastasectomy | 13
Not completed — Other | 71

BASELINE CHARACTERISTICS:
Population: Full analysis population (FAS) included all participants who received bevacizumab in first line mCRC. Baseline characteristics were reported by age groups.
Groups:
- Bevacizumab: Age <70 Years: Participants aged less than (<) 70 years, with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
- Bevacizumab: Age 70-80 Years: Participants aged between 70-80 years, with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
- Bevacizumab: Age >80 Years: Participants aged greater than (>) 80 years, with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab: Age <70 Years | Bevacizumab: Age 70-80 Years | Bevacizumab: Age >80 Years | Total
Number analyzed (Participants) | 120 | 66 | 13 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] — Reported age data represents age at screening; calculated as: (screening date minus [-] birth date) divided by (/) 365.25.
  years | 60.0 (7.7) | 74.3 (2.7) | 83.8 (2.4) | 66.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 32 | 4 | 83
  Male | 73 | 34 | 9 | 116

OUTCOME MEASURES:

1. Primary Outcome: Duration of Bevacizumab Treatment
Description: Duration of bevacizumab treatment (in months) was defined as: (last treatment date - first treatment date plus [+] 1)/30.44. Duration of treatment was estimated using Kaplan-Meier method. Results are reported as per age groups (<70 years and greater than or equal to [≥] 70 years) as well as for overall participants.
Time Frame: Baseline up to end of treatment (up to approximately 3 years)
Population: FAS.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab: Age <70 Years: Participants aged < 70 years, with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
- Bevacizumab: Age ≥70 Years: Participants aged greater than or equal to (≥) 70 years, with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed. Due to the small number of participants aged >80 years, the age groups "70-80 Years" and ">80 Years" have been pooled in this group.
- Bevacizumab: Overall: All participants with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
Arm/Group | Bevacizumab: Age <70 Years | Bevacizumab: Age ≥70 Years | Bevacizumab: Overall
Number analyzed (Participants) | 120 | 79 | 199
months | 6.50 [5.26 to 7.39] | 5.09 [3.48 to 6.24] | 5.95 [5.09 to 6.80]
Statistical Analysis 1: Comparison: Bevacizumab: Age <70 Years vs Bevacizumab: Age ≥70 Years; Test type: Superiority or Other; p = 0.8579, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.70 to 1.54]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS (in months) was defined as: (date of progression or censored date - first date of treatment + 1)/30.44. Date of progression was derived from Response Evaluation Criteria in Solid Tumors (RECIST) evaluation or from last available date for participant who withdrew the study for progressive disease without progression according to RECIST evaluation. Progression was defined (as per RECIST) as at least a 20 percent (%) increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or appearance of one or more new non-target lesions and/or unequivocal progression of existing non-target lesions. PFS was estimated using Kaplan-Meier method. Results are reported as per age groups (<70 years and ≥70 years) as well as for overall participants.
Time Frame: Baseline up to disease progression or death (up to approximately 3 years)
Population: FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: Age <70 Years | Bevacizumab: Age ≥70 Years | Bevacizumab: Overall
Number analyzed (Participants) | 120 | 79 | 199
months | 11.47 [9.72 to 13.63] | 12.68 [7.88 to 19.84] | 11.53 [9.86 to 13.73]
Statistical Analysis 1: Comparison: Bevacizumab: Age <70 Years vs Bevacizumab: Age ≥70 Years; Test type: Superiority or Other; p = 0.1555, Regression, Cox; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.30 to 1.21]

3. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Tumor response was assessed using RECIST. Complete Response (CR): disappearance of all target and non-target lesions; Partial Response (PR): at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions or appearance of one or more new non-target lesions and/or unequivocal progression of existing non-target lesions; Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started or persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits. Results are reported as per age groups (<70 years, 70-80 years, and >80 years) as well as for overall participants.
Time Frame: Baseline up to disease progression or death (up to approximately 3 years)
Population: FAS. Here, number of participants analyzed = participants with available data for this outcome.
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab: Age <70 Years: Participants aged <70 years, with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
- Bevacizumab: Age >80 Years: Participants aged >80 years, with mCRC for whom the physician decided to prescribe bevacizumab as part of their first line treatment and in line with current SmPC (or local label). The decision to prescribe bevacizumab was independent of the study and was the responsibility of the treating physician. All concomitant medications as used in daily routine clinical practice were allowed.
Arm/Group | Bevacizumab: Age <70 Years | Bevacizumab: Age 70-80 Years | Bevacizumab: Age >80 Years | Bevacizumab: Overall
Number analyzed (Participants) | 107 | 58 | 13 | 178
percentage of participants
  CR | 3.7 | 3.4 | 7.7 | 3.9
  PR | 43.9 | 46.6 | 53.8 | 45.5
  SD | 46.7 | 36.2 | 23.1 | 41.6
  PD | 5.6 | 12.1 | 15.4 | 8.4
  Not Evaluable | 0.0 | 1.7 | 0.0 | 0.6

4. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG performance status measured on a 6 point scale to assess participant's performance status. 0=Fully active, able to carry on all pre-disease activities without restriction; 1=Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2=Ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=Capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=Completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=Dead. 0=Best status, 5=Worst status. For each time-point, only categories with available data are reported.
Time Frame: Baseline up to Cycle 51 (1 cycle = 21 days)
Population: FAS. Here, number of participants analyzed = participants with available data for this outcome and n = participants with available data for specified category, for each arm, respectively. No participants were evaluable for Cycles 48-50; hence, no data reported for these cycles.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: Age <70 Years | Bevacizumab: Age 70-80 Years | Bevacizumab: Age >80 Years | Bevacizumab: Overall
Number analyzed (Participants) | 108 | 63 | 9 | 180
percentage of participants
  Baseline: ECOG 0 (n=108,63,9,180) | 47.2 | 41.3 | 22.2 | 43.9
  Baseline: ECOG 1 (n=108,63,9,180) | 44.4 | 46.0 | 77.8 | 46.7
  Baseline: ECOG 2 (n=108,63,9,180) | 6.5 | 11.1 | 0.0 | 7.8
  Baseline: ECOG 3 (n=108,63,9,180) | 0.0 | 1.6 | 0.0 | 0.6
  Baseline: ECOG 4 (n=108,63,9,180) | 1.9 | 0.0 | 0.0 | 1.1
  Cycle 1: ECOG 0 (n=101,58,9,168) | 47.5 | 39.7 | 22.2 | 43.5
  Cycle 1: ECOG 1 (n=101,58,9,168) | 43.6 | 51.7 | 77.8 | 48.2
  Cycle 1: ECOG 2 (n=101,58,9,168) | 8.9 | 6.9 | 0.0 | 7.7
  Cycle 1: ECOG 3 (n=101,58,9,168) | 0.0 | 1.7 | 0.0 | 0.6
  Cycle 2: ECOG 0 (n=98,54,8,160) | 44.9 | 38.9 | 37.5 | 42.5
  Cycle 2: ECOG 1 (n=98,54,8,160) | 46.9 | 50.0 | 62.5 | 48.8
  Cycle 2: ECOG 2 (n=98,54,8,160) | 8.2 | 11.1 | 0.0 | 8.8
  Cycle 3: ECOG 0 (n=94,48,7,149) | 50.0 | 41.7 | 42.9 | 47.0
  Cycle 3: ECOG 1 (n=94,48,7,149) | 44.7 | 47.9 | 57.1 | 46.3
  Cycle 3: ECOG 2 (n=94,48,7,149) | 5.3 | 10.4 | 0.0 | 6.7
  Cycle 4: ECOG 0 (n=87,45,7,139) | 52.9 | 40.0 | 28.6 | 47.5
  Cycle 4: ECOG 1 (n=87,45,7,139) | 43.7 | 46.7 | 71.4 | 46.0
  Cycle 4: ECOG 2 (n=87,45,7,139) | 3.4 | 13.3 | 0.0 | 6.5
  Cycle 5: ECOG 0 (n=88,36,6,130) | 48.9 | 36.1 | 16.7 | 43.8
  Cycle 5: ECOG 1 (n=88,36,6,130) | 47.7 | 52.8 | 66.7 | 50.0
  Cycle 5: ECOG 2 (n=88,36,6,130) | 2.3 | 11.1 | 16.7 | 5.4
  Cycle 5: ECOG 3 (n=88,36,6,130) | 1.1 | 0.0 | 0.0 | 0.0
  Cycle 6: ECOG 0 (n=75,36,5,116) | 50.7 | 36.1 | 20.0 | 44.8
  Cycle 6: ECOG 1 (n=75,36,5,116) | 45.3 | 55.6 | 80.0 | 50.0
  Cycle 6: ECOG 2 (n=75,36,5,116) | 4.0 | 8.3 | 0.0 | 5.2
  Cycle 7: ECOG 0 (n=67,31,6,104) | 52.2 | 48.4 | 33.3 | 50.0
  Cycle 7: ECOG 1 (n=67,31,6,104) | 44.8 | 45.2 | 50.0 | 45.2
  Cycle 7: ECOG 2 (n=67,31,6,104) | 3.0 | 6.5 | 16.7 | 4.8
  Cycle 8: ECOG 0 (n=63,26,5,94) | 55.6 | 34.6 | 20.0 | 47.9
  Cycle 8: ECOG 1 (n=63,26,5,94) | 39.7 | 61.5 | 60.0 | 46.8
  Cycle 8: ECOG 2 (n=63,26,5,94) | 4.8 | 3.8 | 20.0 | 5.3
  Cycle 9: ECOG 0 (n=62,27,4,93) | 50.0 | 44.4 | 25.0 | 47.3
  Cycle 9: ECOG 1 (n=62,27,4,93) | 45.2 | 51.9 | 50.0 | 47.3
  Cycle 9: ECOG 2 (n=62,27,4,93) | 4.8 | 3.7 | 25.0 | 5.4
  Cycle 10: ECOG 0 (n=53,29,3,85) | 56.6 | 51.7 | 0.0 | 52.9
  Cycle 10: ECOG 1 (n=53,29,3,85) | 37.7 | 41.4 | 100.0 | 41.2
  Cycle 10: ECOG 2 (n=53,29,3,85) | 5.7 | 6.9 | 0.0 | 5.9
  Cycle 11: ECOG 0 (n=54,21,4,79) | 57.4 | 42.9 | 25.0 | 51.9
  Cycle 11: ECOG 1 (n=54,21,4,79) | 38.9 | 57.1 | 50.0 | 44.3
  Cycle 11: ECOG 2 (n=54,21,4,79) | 3.7 | 0.0 | 25.0 | 3.8
  Cycle 12: ECOG 0 (n=48,21,3,72) | 58.3 | 47.6 | 0.0 | 52.8
  Cycle 12: ECOG 1 (n=48,21,3,72) | 35.4 | 52.4 | 66.7 | 41.7
  Cycle 12: ECOG 2 (n=48,21,3,72) | 6.3 | 0.0 | 33.3 | 5.6
  Cycle 13: ECOG 0 (n=39,17,1,57) | 53.8 | 41.2 | 0.0 | 49.1
  Cycle 13: ECOG 1 (n=39,17,1,57) | 41.0 | 58.8 | 100.0 | 47.4
  Cycle 13: ECOG 2 (n=39,17,1,57) | 5.1 | 0.0 | 0.0 | 3.5
  Cycle 14: ECOG 0 (n=34,15,1,50) | 50.0 | 40.0 | 0.0 | 46.0
  Cycle 14: ECOG 1 (n=34,15,1,50) | 47.1 | 53.3 | 100.0 | 50.0
  Cycle 14: ECOG 2 (n=34,15,1,50) | 2.9 | 6.7 | 0.0 | 4.0
  Cycle 15: ECOG 0 (n=30,14,1,45) | 60.0 | 42.9 | 0.0 | 53.3
  Cycle 15: ECOG 1 (n=30,14,1,45) | 40.0 | 57.1 | 100.0 | 46.7
  Cycle 16: ECOG 0 (n=28,13,1,42) | 57.1 | 38.5 | 0.0 | 50.0
  Cycle 16: ECOG 1 (n=28,13,1,42) | 42.9 | 61.5 | 100.0 | 50.0
  Cycle 17: ECOG 0 (n=24,11,1,36) | 58.3 | 45.5 | 0.0 | 52.8
  Cycle 17: ECOG 1 (n=24,11,1,36) | 41.7 | 54.5 | 100.0 | 47.2
  Cycle 18: ECOG 0 (n=18,9,1,28) | 50.0 | 22.2 | 0.0 | 39.3
  Cycle 18: ECOG 1 (n=18,9,1,28) | 50.0 | 77.8 | 100.0 | 60.7
  Cycle 19: ECOG 0 (n=19,10,1,30) | 57.9 | 30.0 | 0.0 | 46.7
  Cycle 19: ECOG 1 (n=19,10,1,30) | 42.1 | 70.0 | 100.0 | 53.3
  Cycle 20: ECOG 0 (n=15,6,0,21) | 53.3 | 33.3 | NA — Data not available as no participant was evaluable. | 47.6
  Cycle 20: ECOG 1 (n=15,6,0,21) | 46.7 | 66.7 | NA — Data not available as no participant was evaluable. | 52.4
  Cycle 21: ECOG 0 (n=15,5,0,20) | 73.3 | 0.0 | NA — Data not available as no participant was evaluable. | 55.0
  Cycle 21: ECOG 1 (n=15,5,0,20) | 26.7 | 100.0 | NA — Data not available as no participant was evaluable. | 45.0
  Cycle 22: ECOG 0 (n=16,5,0,21) | 50.0 | 0.0 | NA — Data not available as no participant was evaluable. | 38.1
  Cycle 22: ECOG 1 (n=16,5,0,21) | 50.0 | 100.0 | NA — Data not available as no participant was evaluable. | 61.9
  Cycle 23: ECOG 0 (n=12,5,0,17) | 50.0 | 0.0 | NA — Data not available as no participant was evaluable. | 35.3
  Cycle 23: ECOG 1 (n=12,5,0,17) | 50.0 | 100.0 | NA — Data not available as no participant was evaluable. | 64.7
  Cycle 24: ECOG 0 (n=10,5,0,15) | 70.0 | 20.0 | NA — Data not available as no participant was evaluable. | 53.3
  Cycle 24: ECOG 1 (n=10,5,0,15) | 30.0 | 60.0 | NA — Data not available as no participant was evaluable. | 40.0
  Cycle 24: ECOG 2 (n=10,5,0,15) | 0.0 | 20.0 | NA — Data not available as no participant was evaluable. | 6.7
  Cycle 25: ECOG 0 (n=9,4,0,13) | 77.8 | 0.0 | NA — Data not available as no participant was evaluable. | 53.8
  Cycle 25: ECOG 1 (n=9,4,0,13) | 22.2 | 100.0 | NA — Data not available as no participant was evaluable. | 46.2
  Cycle 26: ECOG 0 (n=9,4,0,13) | 77.8 | 25.0 | NA — Data not available as no participant was evaluable. | 61.5
  Cycle 26: ECOG 1 (n=9,4,0,13) | 22.2 | 75.0 | NA — Data not available as no participant was evaluable. | 38.5
  Cycle 27: ECOG 0 (n=8,4,0,12) | 100.0 | 0.0 | NA — Data not available as no participant was evaluable. | 66.7
  Cycle 27: ECOG 1 (n=8,4,0,12) | 0.0 | 100.0 | NA — Data not available as no participant was evaluable. | 33.3
  Cycle 28: ECOG 0 (n=5,4,0,9) | 80.0 | 0.0 | NA — Data not available as no participant was evaluable. | 44.4
  Cycle 28: ECOG 1 (n=5,4,0,9) | 20.0 | 100.0 | NA — Data not available as no participant was evaluable. | 55.6
  Cycle 29: ECOG 0 (n=6,4,0,10) | 83.3 | 0.0 | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 29: ECOG 1 (n=6,4,0,10) | 16.7 | 75.0 | NA — Data not available as no participant was evaluable. | 40.0
  Cycle 29: ECOG 2 (n=6,4,0,10) | 0.0 | 25.0 | NA — Data not available as no participant was evaluable. | 10.0
  Cycle 30: ECOG 0 (n=6,4,0,10) | 83.3 | 0.0 | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 30: ECOG 1 (n=6,4,0,10) | 16.7 | 75.0 | NA — Data not available as no participant was evaluable. | 40.0
  Cycle 30: ECOG 2 (n=6,4,0,10) | 0.0 | 25.0 | NA — Data not available as no participant was evaluable. | 10.0
  Cycle 31: ECOG 0 (n=6,3,0,9) | 83.3 | 0.0 | NA — Data not available as no participant was evaluable. | 55.6
  Cycle 31: ECOG 1 (n=6,3,0,9) | 16.7 | 100.0 | NA — Data not available as no participant was evaluable. | 44.4
  Cycle 32: ECOG 0 (n=5,3,0,8) | 100.0 | 0.0 | NA — Data not available as no participant was evaluable. | 62.5
  Cycle 32: ECOG 1 (n=5,3,0,8) | 0.0 | 100.0 | NA — Data not available as no participant was evaluable. | 37.5
  Cycle 33: ECOG 0 (n=6,3,0,9) | 100.0 | 0.0 | NA — Data not available as no participant was evaluable. | 66.7
  Cycle 33: ECOG 1 (n=6,3,0,9) | 0.0 | 100.0 | NA — Data not available as no participant was evaluable. | 33.3
  Cycle 34: ECOG 0 (n=5,3,0,8) | 80.0 | 0.0 | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 34: ECOG 1 (n=5,3,0,8) | 0.0 | 100.0 | NA — Data not available as no participant was evaluable. | 37.5
  Cycle 34: ECOG 2 (n=5,3,0,8) | 20.0 | 0.0 | NA — Data not available as no participant was evaluable. | 12.5
  Cycle 35: ECOG 0 (n=5,2,0,7) | 60.0 | 0.0 | NA — Data not available as no participant was evaluable. | 42.9
  Cycle 35: ECOG 1 (n=5,2,0,7) | 20.0 | 100.0 | NA — Data not available as no participant was evaluable. | 42.9
  Cycle 35: ECOG 2 (n=5,2,0,7) | 20.0 | 0.0 | NA — Data not available as no participant was evaluable. | 14.3
  Cycle 36: ECOG 0 (n=5,2,0,7) | 60.0 | 0.0 | NA — Data not available as no participant was evaluable. | 42.9
  Cycle 36: ECOG 1 (n=5,2,0,7) | 20.0 | 100.0 | NA — Data not available as no participant was evaluable. | 42.9
  Cycle 36: ECOG 2 (n=5,2,0,7) | 20.0 | 0.0 | NA — Data not available as no participant was evaluable. | 14.3
  Cycle 37: ECOG 0 (n=5,1,0,6) | 60.0 | 0.0 | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 37: ECOG 1 (n=5,1,0,6) | 20.0 | 100.0 | NA — Data not available as no participant was evaluable. | 33.3
  Cycle 37: ECOG 2 (n=5,1,0,6) | 20.0 | 0.0 | NA — Data not available as no participant was evaluable. | 16.7
  Cycle 38: ECOG 0 (n=5,1,0,6) | 60.0 | 0.0 | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 38: ECOG 1 (n=5,1,0,6) | 20.0 | 100.0 | NA — Data not available as no participant was evaluable. | 33.3
  Cycle 38: ECOG 2 (n=5,1,0,6) | 20.0 | 0.0 | NA — Data not available as no participant was evaluable. | 16.7
  Cycle 39: ECOG 0 (n=4,1,0,5) | 50.0 | 0.0 | NA — Data not available as no participant was evaluable. | 40.0
  Cycle 39: ECOG 1 (n=4,1,0,5) | 25.0 | 100.0 | NA — Data not available as no participant was evaluable. | 40.0
  Cycle 39: ECOG 2 (n=4,1,0,5) | 25.0 | 0.0 | NA — Data not available as no participant was evaluable. | 20.0
  Cycle 40: ECOG 0 (n=3,1,0,4) | 66.7 | 0.0 | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 40: ECOG 1 (n=3,1,0,4) | 0.0 | 100.0 | NA — Data not available as no participant was evaluable. | 25.0
  Cycle 40: ECOG 2 (n=3,1,0,4) | 33.3 | 0.0 | NA — Data not available as no participant was evaluable. | 25.0
  Cycle 41: ECOG 0 (n=2,0,0,2) | 50.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 41: ECOG 2 (n=2,0,0,2) | 50.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 42: ECOG 0 (n=3,0,0,3) | 33.3 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 33.3
  Cycle 42: ECOG 1 (n=3,0,0,3) | 33.3 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 33.3
  Cycle 42: ECOG 2 (n=3,0,0,3) | 33.3 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 33.3
  Cycle 43: ECOG 0 (n=2,0,0,2) | 50.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 43: ECOG 2 (n=2,0,0,2) | 50.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 44: ECOG 0 (n=2,0,0,2) | 50.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 50.0
  Cycle 44: ECOG 2 (n=2,0,0,2) | 50.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 50.0
  Cycles 45: ECOG 2 (n=1,0,0,1) | 100.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 100.0
  Cycles 46: ECOG 2 (n=1,0,0,1) | 100.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 100.0
  Cycles 47: ECOG 2 (n=1,0,0,1) | 100.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 100.0
  Cycles 51: ECOG 1 (n=1,0,0,1) | 100.0 | NA — Data not available as no participant was evaluable. | NA — Data not available as no participant was evaluable. | 100.0

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Arm/Group | Bevacizumab: Overall
Serious Adverse Events (participants affected / at risk) | 94/201
Other Adverse Events (participants affected / at risk) | 34/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab: Overall (N=201)
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Agranulocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Granulocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 15
Large intestine perforation (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 5
Enteritis (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Dyschezia (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Anal Fissure (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1
Faecalith (Gastrointestinal disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 10
Inflammation (General disorders) | 1
Pain (General disorders) | 2
Disease progression (General disorders) | 3
Fatigue (General disorders) | 2
Asthenia (General disorders) | 3
Mucosal inflammation (General disorders) | 4
General physical health deterioration (General disorders) | 6
Chest pain (General disorders) | 1
Unevaluable event (General disorders) | 1
Ulcer (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 2
Portal vein thrombosis (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Bacterial prostatitis (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 3
Anal abscess (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 3
Colonic abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Spinal cord infection (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pelvic abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
General physical condition abnormal (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Epilepsy (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Peripheral paralysis (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Cancer surgery (Surgical and medical procedures) | 2
Hepatectomy (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 2
Venous thrombosis (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab: Overall (N=201)
Neutropenia (Blood and lymphatic system disorders) | 14
Anaemia (Blood and lymphatic system disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 31
Abdominal pain (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 22
Decreased appetite (Metabolism and nutrition disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.